CLINICAL TRIAL: NCT02465424
Title: Assessing Quality of Life Tools in Medullary Thyroid Cancer Patients
Acronym: QaLM
Status: Completed | Type: Observational
Sponsor: Velindre NHS Trust (Other Government)
Responsible Party: Principal Investigator, Dr Laura Moss, Consultant Clinical Oncologist, Velindre NHS Trust
Other Study IDs: QaLM
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Medullary Thyroid Cancer
Keywords: quality of life questionnaires
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- questionnaire order: the order of presentation of the 4 quality of life questionnaires to the patients will be randomised to reduce the impact of boredom and habituation on responses
  Interventions: Other: quality of life questionnaires

INTERVENTIONS:
Other: quality of life questionnaires — Randomised allocation of 4 validated quality of life questionnaires followed by study specific overview questionnaire
  Other Names: health related quality of life tools

SUMMARY:
The purpose of this study is to determine which Health Related Quality of Life (HRQoL) tools patients with medullary thyroid cancer (MTC) find most helpful. The study will compare a generic cancer QoL tool with those developed for thyroid cancer patients and neuroendocrine tumour (NET) patients. The study will also evaluate clinicians' opinions on the clinical usefulness of the QoL tools.

DETAILED DESCRIPTION:
Background Currently available thyroid cancer quality of life (QoL) tools tend to be focused on issues more relevant to patients with differentiated thyroid cancer (DTC) rather than medullary thyroid cancer (MTC). As MTC is a neuroendocrine tumour (NET) patients often have symptoms more in common with patients with these types of tumours rather than patients with other types of thyroid cancer.

MTC presents as a sporadic tumour in approximately 75% of cases and as an inherited disease in 25%. The inherited forms of MTC constitute part of the Multiple Endocrine Neoplasia disorders. Patients with Multiple Endocrine Neoplasia (MEN) may therefore have a number of medical conditions which can impact on their quality of life.

Patients with rare diseases can face additional barriers and concerns such as limited patient information resources, the potential for lack of understanding amongst family and friends and they will inevitably encounter healthcare professionals who do not have experience of managing their rare condition.

It can be difficult to fully appreciate the impact of a cancer diagnosis or an inherited syndrome, raised and rising tumour markers and disease symptoms on a patient's quality of life.

Quality of life is multi faceted and is affected by emotional, social and functional issues as well as disease related problems. Quality of life tools can increase the information a healthcare professional obtains about a patient thus facilitating the consultation as well as improving the patient's satisfaction with the consultation.

Patients with raised or rising tumour markers (calcitonin and carcinoembryonic antigen (CEA)) often remain physically well and of good performance status but there can be a significant amount of distress associated with the awareness of abnormal or worsening biochemical results.

Once MTC has spread beyond the neck, curative options are lacking and the aim of treatment switches to maintenance of quality of life and palliation of symptoms. Therapeutic interventions may include somatostatin analogue therapy, radiolabelled therapy such as mIBG therapy or targeted therapy using tyrosine kinase inhibitors such as vandetanib and cabozantinib. It can be difficult to decide when to start systemic targeted therapy as the drugs themselves can have significant toxicities which can impact on quality of life and they have only been shown to achieve a modest increase in progression free survival and not overall survival. These agents are taken orally on a daily basis and treatment can extend for years in some cases. If the investigators had a robust tool to assess MTC related QOL clinicians may find it easier to select those patients who will benefit most from systemic anti cancer therapies as opposed to more simple supportive symptomatic measures.

Aims

The aim of the study is to determine which Health Related Quality of Life (HRQoL) instruments patients with sporadic and inherited MTC and early and advanced stage medullary thyroid cancer patients find most helpful in facilitating communication of their health problems to their clinicians. The study will attempt to ascertain if this patient cohort's symptoms and quality of life is better assessed by a thyroid cancer specific questionnaire, a general symptom questionnaire or a neuroendocrine tumour specific questionnaire.

The study will also ascertain clinician's views on the quality of life tools in terms of their ability to highlight problems not otherwise ascertained by a standard clinical review appointment along with the relationship between quality of life tool score, performance status and disease burden.

Trial Design

Patients will be randomised to complete four quality of life questionnaires in different sequences and then will be asked questions about which questionnaire they prefer in a final brief questionnaire.

The questionnaires will be presented to the participant in random order to counterbalance the effects of boredom and habituation. A trained nurse or researcher will be available to assist with the completion of the questionnaires when required.

A small cohort of study participants (approx 10-15) will undergo cognitive interviews. This will help test the functionality of the survey questions. The interviews will take the format of retrospective probes i.e. directed questions undertaken by a member of the research team after the participant has completed all the questionnaires. The aim is identify problems not covered by the questionnaires, problems with terminology and comprehension as well as assessing the ability of the participants to successfully rank the 4 quality of life tools.

Outcomes

o Primary outcome measure: Identification of medullary thyroid cancer patients' preferred quality of life instrument for describing their concerns and for facilitating communication with their health care professional. Assessed by patients' ranking of the questionnaires from 1-4 (with 1 representing the most favoured tool).

* Secondary Outcomes:
* assess if there are differences between preferred quality of life tools amongst sporadic and inherited MTC patients
* correlate quality of life questionnaire scores with performance status, disease stage and burden, calcitonin doubling time
* assess clinicians' views on the quality of life tools in terms of their ability to highlight problems not otherwise ascertained by a standard clinical review appointment

Eligibility: 200 patients required

* Patients 16 years old or over who have a diagnosis of medullary thyroid cancer (inherited or sporadic)
* Patients can be included at any time point after diagnosis

Exclusion Criteria:

* Patients who have differentiated (papillary or follicular) thyroid cancer or anaplastic thyroid cancer or lymphoma of the thyroid.
* Patients who do not sufficiently understand the English language or patients with learning disabilities, as these are standardised and validated questionnaires that are in English.

Quality of Life Questionnaires

The study will utilise both generic quality of life instruments as well as disease specific ones. The generic instrument will be EORTC QLQ-C30 and the disease specific tools will be the MD Anderson Symptom Inventory (MDASI) thyroid module and the City of Hope Quality of Life Scale/THYROID (amended) which assess thyroid cancer issues and EORTC QLQ-GINET21 which assesses issues relevant to neuroendocrine tumours.

i) EORTC QLQ-C30 core quality of life questionnaire is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items. It focuses on the QoL consequences of physical limitations and on clinical symptoms. It is a generic measure, as opposed to one that targets a specific disease.

ii) MD Anderson Symptom Inventory (MDASI) thyroid module is a patient reported outcome measure that assesses the severity of multiple symptoms and the impact of symptoms on daily functioning during the last 24 hours. The 1-10 point rating scale is comprised of the 13 core items, 6 thyroid specific symptoms and 5 psychosocial items. Completion of the measure is simple and takes only a few minutes.

iii) The City of Hope Quality of Life Scale/THYROID (amended) Questions relate to specific issues of concern to thyroid patients regarding the condition itself, treatment and side effects. Items cover physical, psychological, social and spiritual domains. It is an established instrument specifically designed for use with thyroid patients. The original tool used some questions relevant to differentiated thyroid cancer treatment which are not relevant to MTC patients so these have been substituted for questions specific to the management of MTC. These amendments are not therefore part of the validated tool but are believed to be important and relevant to this study.

iv) EORTC QLQ-GINET21This has been reported to be a responsive tool for assessing quality of life for neuroendocrine tumours arising in the gastrointestinal tract, pancreas and liver. A significant proportion of patients with advanced medullary thyroid cancer experience gastrointestinal symptoms related to hypercalcitoninaemia so this study is an opportunity to assess if this QOL tool is relevant and helpful in describing quality of life concerns for MTC patients who have a different form of neuroendocrine tumour.

Patients Preference

After completing each of the four questionnaires, patients are asked to answer a few additional brief questions to assess whether they found that particular questionnaire useful, as well as questions regarding questionnaire characteristics (length, ease of understanding and relevance to health problems). There is also a free text area for comments on areas patients may consider important but which are not covered by the questionnaires. After completing all 4 questionnaires patients are asked to evaluate all of the quality of life tools in a final short series of questions and to rank the QoL tools in order, 1-4, with 1 being the QoL tool they found most helpful and 4 for the QoL tool which was least helpful.

Publication

The results of the trial will be shared with the clinical community via publications in peer-reviewed journals and presentations at national/international meetings.

Any publications or presentations arising directly as a result of this project will acknowledge all contributing investigators and funders.

Study Support

The QaLM protocol has been reviewed by members of the NCRI Thyroid Cancer Subgroup, Thyroid Cancer Support Group Wales, Butterfly Thyroid Cancer Trust and AMEND. Widespread support has been expressed from clinicians and patient representatives alike and to date 16 leading UK thyroid cancer teams have expressed interest in participating in the study.

It is anticipated that the QaLM study would be eligible for inclusion in the National Cancer Research Institute's (NCRI) Thyroid Cancer Trial portfolio which would facilitate the multicentre participation and recruitment required for successful completion of the study.

The study proposal was presented at a NCRI Thyroid Cancer Subgroup research meeting in October 2014 and leading UK clinicians requested that the number of patients recruited be increased from 100 to 200 to take in to account the unique opportunity to offer a study to this patient group.

Biochemical monitoring (calcitonin and CEA) forms a routine part of the investigation and follow up of patients with medullary thyroid cancer and it is known that the rate of change in biochemical markers can predict likely survival. It is not known however if there is any association between biochemical marker changes and quality of life. This project would be a unique opportunity to compare and contrast issues faced by patients with MTC arising as part of Multiple Endocrine Neoplasia and those where MTC arises sporadically.

In the era of new systemic therapies in the form of oral tyrosine kinase inhibitor drugs, that are potentially taken long term, require frequent monitoring when initiated and have significant potential toxicities, it would be beneficial to try and quantify and compare the problems caused by the disease and those caused by systemic therapy. Quality of life is paramount and the investigators currently lack information on the burden of disease and treatment. This information could help commissioners appraise new therapies and be used alongside clinical and cost effectiveness data.

ELIGIBILITY:
Inclusion Criteria:

* Patients 16 years old or over who have a diagnosis of medullary thyroid cancer (inherited or sporadic)
* Patients can be included at any time point after diagnosis

Exclusion Criteria:

* Patients who have differentiated (papillary or follicular) thyroid cancer or anaplastic thyroid cancer or lymphoma of the thyroid.
* Patients who do not sufficiently understand the English language or patients with learning disabilities, as these are standardised and validated questionnaires that are in English.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medullary thyroid cancer patients who are attending a thyroid cancer clinic in tertiary care setting in the NHS
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Ranking of quality of life assessment tool by patients | At recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Laura Moss, MB BCh, Principal Investigator — Velindre NHS Trust
Locations (7):
- United Kingdom (7):
  - Velindre Hospital, Cardiff
  - University Hospitals of Coventry and Warwickshire, Coventry
  - Western general Hospital, Edinburgh
  - Imperial Hospital, London
  - St. Bartholomew's Hospital, London
  - Christie Hospital, Manchester
  - Weston Park Hospital, Sheffield